CLINICAL TRIAL: NCT00029991
Title: Extract of Ginkgo Biloba (Egb 761) and Vascular Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AT000204-02 (NIH)
Record Dates: First submitted 2002-01-29; First posted 2002-01-30 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease
Keywords: Leg pain; Peripheral angiopathies; Vascular Diseases, peripheral
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases | interventions — Ginkgo Extract

INTERVENTIONS:
Drug: Gingko Biloba (Herb)

SUMMARY:
This study will determine if a highly standardized herbal extract of the leaves of the Ginkgo Biloba tree will benefit patients who have pain on walking due to narrowing of the arteries of the legs.

DETAILED DESCRIPTION:
This study will determine if a highly standardized herbal extract of the leaves of the Ginkgo Biloba tree, widely used in Europe for two decades, will benefit patients who have pain on walking due to narrowing of the arteries of the legs. A few studies done about ten years ago in Germany appeared to benefit such patients. It is important to confirm these findings and to learn how it may work. Animal studies suggest that this extract, known as EGb 761, works through very strong antioxidant mechanisms. A second action suggested is that it stimulates cells lining the inside of the arteries to produce the compound nitric oxide. These cells, known as endothelial cells, are susceptible to damage by blood cholesterol, smoking or high blood pressure and, when damaged, will allow cholesterol to deposit in arteries. Antioxidants can prevent the endothelial cell damage, therefore it is very important to know if EGb 761 works through that mechanism. These cells also produce nitric oxide naturally as a defense against injury, so an EGb 761 effect on nitric oxide would also provide benefit. Consumption of Gingko Biloba products, many of uncertain purity, is increasing rapidly in the United States. Confirmation of its benefits, derived largely from Europe, is important to protect the health of the American people and to find new and inexpensive remedies for common problems, such as narrowed arteries in the legs. If benefit is found for this problem, then it will be highly likely that the atherosclerotic deposits that cause heart attacks and many strokes may also be preventable or treatable with this compound. Any benefit found will also lead to future studies to determine which constituents of the mixture now present in EGb 761 confers the benefit. If these actions, or others, were discovered, then this herbal product could become used with greater confidence.

This double-blind study will randomly assign parcicipants to receive 4 months of either EGb 761 at 320 mg/day or placebo. Improving walking distances by 30% or greater is the major goal. A second goal will test the safety of EGb 761 through careful examination of liver and kidney function and other measures of general health. Also, a thorough search will occur for antioxidant actions and for changes in endothelial cell nitric oxide production. Two study visits will occur at baseline, and two will occur at Month 4.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females.
* Intermittent claudication or rest pain due to peripheral arterial disease, in a steady clinical state for at least three months according to physician's opinion. The peripheral arterial disease must be confirmed by Doppler ankle brachial index (ABI).
* Wash-out of disallowed medications of at least four weeks prior to screening.
* Patient understands all elements of informed consent and has agreed to it in writing prior to enrollment.

Exclusion Criteria

* Peripheral arterial disease of non-atherosclerotic nature.
* Inability to walk at least 50 feet on a standardized treadmill.
* Any type of major surgery during the last three months and, in particular, aortic or lower extremity arterial surgery, angioplasty, or lumbar sympathectomy within 3 months; leg amputation above the ankle.
* Any disease process, other than PAD, limiting exercise capacity on the treadmill.
* Myocardial infarction in the previous 3 months.
* Current enrollment in another clinical trial and/or ingestion of another investigational product within the past 30 days.
* Diabetes retinopathy, age-related maculopathy, or any other proliferative retinopathy.
* Active malignant disease or history of malignancy.
* Intolerance to sublingual nitroglycerin.
* Uncontrolled hypertension.
* Type I diabetes.
* Use of pentoxifylline, carnitine, arginine or prostacyclin.
* Use of antioxidants other than those in the usual multivitamin mixture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2000-09; Study Completion 2005-07

PRIMARY OUTCOMES:
Maximal and pain-free walking distance

SECONDARY OUTCOMES:
Flow mediated vasodilation of the brachial artery
Antibodies to epitopes of oxidized LDL

CONTACTS AND LOCATIONS:
Overall Officials: John W. Farquhar, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Derived] Gardner CD, Taylor-Piliae RE, Kiazand A, Nicholus J, Rigby AJ, Farquhar JW. Effect of Ginkgo biloba (EGb 761) on treadmill walking time among adults with peripheral artery disease: a randomized clinical trial. J Cardiopulm Rehabil Prev. 2008 Jul-Aug;28(4):258-65. doi: 10.1097/01.HCR.0000327184.51992.b8. PMID 18628657